CLINICAL TRIAL: NCT01425580
Title: Effects on Subclinical Heart Failure in Type 2 Diabetic Subjects on Liraglutide Treatment Versus Glimepiride Both in Combination With Metformin
Brief Title: Liraglutide and Heart Failure in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Nystrom (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Sponsor-Investigator, Thomas Nystrom, MD, PhD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU-nr 2010-022695-31; 2010-022695-31 (EudraCT Number)
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Congestive Heart Failure; Type 2 Diabetes Mellitus
Keywords: Congestive Heart Failure; Type 2 Diabetes Mellitus; GLP-1; Liraglutide
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2 | interventions — Liraglutide; glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- liraglutide (Experimental): The present trial is a two centre, open, assessor-blinded and active-controlled, parallel-group trial, in combination with metformin. The trial will compare the treatment with liraglutide 1.8 mg (s.c) QD + metformin up to 1 g BID, with that of glimepiride 4 mg QD (comparator) + metformin up to 1 g BID, on LV function in subjects with type 2 diabetes.
  Interventions: Drug: liraglutide; Drug: glimepiride; Drug: Metformin
- glimepiride (Active Comparator): 4 mg p.o. (QD)
  Interventions: Drug: liraglutide; Drug: glimepiride; Drug: Metformin

INTERVENTIONS:
Drug: liraglutide — 1.8 mg s.c. (QD)
Drug: glimepiride — 4 mg p.o. (QD)
Drug: Metformin — 500 mg p.o. (BID)

SUMMARY:
Glucagon-like peptide-1 (GLP-1) is a naturally occurring incretin with insulinotropic properties. Apart from the glycemic actions, cardiovascular effects by GLP-1 have recently been reviewed. Receptors for GLP-1 are expressed in the rodent and human heart and acute activation of GLP-1 signalling has been shown to influence e.g. heart rate and blood pressure. In a knock-out mouse model, GLP-1R-/- mice exhibited a defective cardiovascular contractile response together with left ventricular hypertrophy. GLP-1 improves severe left ventricular heart failure in humans suffering from a myocardial infarction. Hence, it has been demonstrated that GLP-1 exerts direct functional effects through both GLP-1 receptor dependent and independent pathways in the heart.

Native GLP-1 is an extremely short acting peptide, with a half-time breakdown of 1-2 minutes, a feature that makes it unsuitable as a drug treatment for type 2 diabetes. To this end, several long-acting GLP-1 analogues, drugs for treating type 2 diabetes, have been tested for this purpose. The analogue liraglutide exerts its effects via the native GLP-1 receptor, localized not only on the pancreatic β-cells, but also in the human heart. Interestingly, liraglutide has been demonstrated to have beneficial effect on heart function in mice. Taken together, recent data shows that GLP-1 and its stable analogue liraglutide exert beneficial cardiovascular effects.

The purpose of this study is to determine whether the glucagon-like peptide-1 (GLP-1) analogue liraglutide improves heart function (measured as left ventricle longitudinal function and/or functional reserve during rest and/or after exercise) after 18 weeks of liraglutide + metformin, compared with glimepiride + metformin, using tissue Doppler echocardiography.

DETAILED DESCRIPTION:
The subjects will attend a screening visit (Visit 1) in order to assess their eligibility. If found eligible, the subjects will return at Visit 2 within approximately 4 weeks, after Visit 1, with an up-titration with metformin 1 g BID or the maximal tolerated dosage of metformin (Run-in period).

At Visit 2 patients will be tested for;

* Heart function at rest and during an exercise ECG Stress Test with tissue Doppler echocardiography
* 24-hour blood pressure
* Anthropometric assessment
* Symptoms of dyspnea or fatigue (scoring system, classified as NYHA).
* Quality of life (SF 36)
* Blood test (venipuncture)

Subsequently thereafter, subjects will during visit 2 be randomized to receive either liraglutide 1.8 mg s.c. (initial dose of 0.6 mg with an up-titration of 0.6 mg every week, final dose 1.8 mg QD) or glimepiride 4 mg p.o (initial dose of 2 mg, with an up-titration of 1 mg every week, final dose 4 mg QD).

At Visit 2, subjects will be supplied with a glucose meter (Abbot Contour) and instruction on use of the device including regular calibration according to the manufacturer's instruction. Subjects will be instructed on how to record the results of the self measured plasma glucose (SMPG) values in the meter. Subjects will then ask to monitor a 7 point profile glucose curve consecutively in three days before visit 3, at visit 4 and at the end of treatment (visit 5). SMBG values will be transferred via a computerized system (Diasend®).

Visit 3. Telephone visit. Self-reporting glucose measurements.

Visit 4. Telephone visit. Self-reporting glucose measurements.

At week 18 (Visit 5), subjects will be re-tested for:

* Heart function at rest and during an exercise ECG Stress Test with tissue Doppler echocardiography
* 24-hour blood pressure
* Anthropometric assessment
* Symptoms of dyspnea or fatigue (scoring system, classified as NYHA).
* Quality of life (SF 36)
* Blood test (venipuncture)

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes.
2. Heart Failure, visualized with echocardiography, one of the following (2.1, 2.2 or 2.3).

   * Ejection Fraction ≤ 50%.
   * Decreased systolic velocity (four chamber view) where two, out of four segments (Septum, Lateral, Inferior and Anterior Wall) has a relative decrease in velocity of 20% compared to a normal population.
   * Evidence of diastolic dysfunction as shown by abnormal left ventricular relaxation, filling, diastolic distensibility or stiffness. An E/E' ratio (ratio of early diastolic velocities of mitral inflow derived Doppler imaging and myocardial movement derived by tissue Doppler imaging) >15 is considered diagnostic of diastolic dysfunction and an E/E' ratio < 8 as diagnostic of the absence of diastolic heart failure. An increased left atrial size (>49 ml/ m2) and an increased left ventricular mass (>122 g/m2 in women and >149 g/m2 in men) are considered sufficient evidence of diastolic dysfunction when the E/E' ratio is inconclusive.
3. HbA1c (accordingly to IFCC) 47 mmol/mol - 95 mmol/mol.
4. If antihypertensive treatment, the medication has to be stable, no change, for the last 1 month.
5. Male and female subjects, 18-80 years of age.
6. Signed informed consent form.

Exclusion Criteria:

1. Type 1 diabetes (autoantibody positive).
2. Any history of receiving GLP-1 analogues or dipeptidyl peptidase inhibitors (DPP-IV inhibitor) or glimeperide.
3. Previous treatment with glitazones within 6 months.
4. Previous treatment with other sulphonylurea within 3 months.
5. Previous treatment with insulin (any regimen) within 1 month.
6. Known severe heart failure, classified as NYHA 3-4.
7. Significant ischemic heart disease (defined as angina-limited exercise or unstable angina); documented acute myocardial infarction (MI) within the previous 8 weeks.
8. Active myocarditis; malfunctioning artificial heart valve.
9. Atria fibrillation or flutter
10. History of ventricular tachycardia within 3 months before study entry; second- or third-degree atrioventricular block.
11. Implanted pacemaker.
12. Supine systolic blood pressure <85 mm Hg or >200 mm Hg.
13. Primary renal impairment (creatinine clearance < 30 ml/min), or creatinine clearance < 60 ml/min if treated with metformin.
14. Uncorrected hypokalemia or hyperkalemia (potassium <3.5 mmol/l or >5.5 mmol/l).
15. Significant anemia (Hb < 90 g/l)
16. Treatment with another investigational agent within 30 days before study entry, judged by the investigator.
17. Severe gastrointestinal disease, including gastroparesis. As judged by the investigator.
18. Body mass index (BMI) > 40 kg/m2.
19. Malignant neoplasm requiring chemotherapy, surgery, radiation or palliative therapy in the previous 5 years. Patients with intraepithelial squamous cell carcinoma of the skin treated with topical 5FU and subjects with basal cell skin cancer are allowed to enter the trial.
20. Females of child bearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice).
21. Current drug and alcohol abuse.
22. History of acute or chronic pancreatitis
23. Subjects considered by the investigator to be unsuitable for the study.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Left ventricle longitudinal function and/or functional reserve during rest and/or after exercise using tissue Doppler echocardiography | 18 weeks

SECONDARY OUTCOMES:
24-hour blood pressure | 18 weeks
Energy delivering from the carotid artery | 18 weeks
N-terminal pro b-type natriuretic peptide (NT-proBNP) levels in serum over time and symptoms of dyspnea or fatigue as assessed by patient and clinician using established scoring systems | 18 weeks
Gene and protein expression (Affymetrix/proteomics) | 18 weeks
Plasma markers of inflammation i.e. hsCRP, IL-6, TNF-α and PAI-1 | 18 weeks
Plasma markers of endothelial activation i.e. E-selectin, VCAM-1, ICAM-1 and plasma levels of nitrate/nitrite | 18 weeks
Lipids | 18 weeks
A1c | 18 week
Body weight | 18 weeks
Adverse events in terms of hypoglycaemia | 18 weeks
Quality of life (SF 36) | 18 weeks
Exercise ECG, including working capacity | 18 weeks
Global LV function (echocardiography) expressed as ejection fraction (EF) | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johan Jendle, MD, PhD, Principal Investigator — University of Örebro
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Department of Clinical Science and Education, Södersjukhuset, Stockholm
  - Karolinska Institutet, Division of Internal Medicine Södersjukhuset AB, Stockholm

REFERENCES:
- [Derived] Scherbak NN, Kruse R, Nystrom T, Jendle J. Glimepiride Compared to Liraglutide Increases Plasma Levels of miR-206, miR-182-5p, and miR-766-3p in Type 2 Diabetes Mellitus: A Randomized Controlled Trial. Diabetes Metab J. 2023 Sep;47(5):668-681. doi: 10.4093/dmj.2022.0342. Epub 2023 Jun 22. PMID 37349083
- [Derived] Jendle J, Hyotylainen T, Oresic M, Nystrom T. Pharmacometabolomic profiles in type 2 diabetic subjects treated with liraglutide or glimepiride. Cardiovasc Diabetol. 2021 Dec 17;20(1):237. doi: 10.1186/s12933-021-01431-2. PMID 34920733
- [Derived] Jendle J, Fang X, Cao Y, Bojo L, Nilsson BK, Hedberg F, Santos-Pardo I, Nystrom T. Effects on repetitive 24-hour ambulatory blood pressure in subjects with type II diabetes randomized to liraglutide or glimepiride treatment both in combination with metformin: a randomized open parallel-group study. J Am Soc Hypertens. 2018 May;12(5):346-355. doi: 10.1016/j.jash.2018.02.003. Epub 2018 Feb 16. PMID 29548934